CLINICAL TRIAL: NCT07011433
Title: Prognostic Value of Pneumonia Pathogens' Virulence Factors and Patient Inflammatory Markers, and Their Associations With Disease Course and Outcome
Brief Title: Pneumonia Pathogens' Virulence Factors, Patient Inflammatory Markers, and Their Associations With Outcomes
Acronym: Pneumonia-1
Status: Enrolling by invitation | Type: Observational
Sponsor: Ruta Nutautiene (Other)
Responsible Party: Sponsor-Investigator, Ruta Nutautiene, PhD Candidate, Pulmonologist, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: 2024-BE10-0003
Record Dates: First submitted 2025-05-07; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Community Acquired Pneumonia (CAP); Hospital Acquired Pneumonia
Keywords: Community-Acquired Pneumonia; Inflammatory Biomarkers; Immune response; Bronchoalveolar Lavage; Procalcitonin
MeSH Terms: conditions — Community-Acquired Pneumonia; Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be retained, however, DNA will not be extracted in the future.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standard Care Group: Participants receive standard pneumonia diagnostics and treatment according to national clinical guidelines, without additional evaluation of immune response biomarkers.
  Interventions: Diagnostic Test: Inflammatory Biomarker Evaluation

INTERVENTIONS:
Diagnostic Test: Inflammatory Biomarker Evaluation — Venous blood samples are collected from subjects and analyzed for inflammatory biomarkers, including CD64, presepsin, IL-6, and IL-8, using a Luminex multiplex assay. Results are used for research purposes only and do not affect clinical management.

SUMMARY:
The study aims to evaluate pneumonia symptoms using physical examinations, radiological and laboratory tests, and prognostic scales such as the Pneumonia Severity Index (PSI) and CURB65. These methods will be combined with the assessment of biomarkers and inflammatory cytokines to enhance clinical decision-making and predict adverse outcomes. Procalcitonin (PCT) levels will help guide the initiation and duration of antibiotic therapy, while variations in treatment may be based on initial levels of inflammatory biomarkers. A notable focus is placed on the CD64 marker, which can increase significantly under the influence of pro-inflammatory cytokines (IL-6, G-CSF) within hours and return to baseline as the infection subsides.

Microbiological testing will be performed selectively, particularly when results could affect antimicrobial therapy choices. Sputum microscopy is planned before antibiotic prescription, with only high-quality samples being considered. Poor-quality sputum will not be further tested. Invasive diagnostic methods will be used only as specified by pneumonia treatment protocols. Bronchoscopy, including bronchoalveolar lavage (BAL), is reserved for severe pneumonia cases under specific conditions, such as failure to expectorate sputum, multiple Gram-negative or fungal isolates, or poor treatment response.

Radiological diagnostics will include chest X-rays in anteroposterior and lateral views, as infiltrates in certain lung segments may be missed on single views. Early radiographic findings may reveal only subtle changes in the lung pattern, so follow-up imaging is planned to ensure an accurate diagnosis. The study will be conducted exclusively in specialized hospital units to maintain patient safety. The collected data will allow for the analysis of relationships between pathogens, their virulence, immune responses, and disease outcomes.

DETAILED DESCRIPTION:
The study will assess pneumonia symptoms based on physical examination and additional data (radiological or laboratory tests), supported by prognostic scales such as the Pneumonia Severity Index (PSI), CURB65 (Annexes No. 7 and 8), in combination with biomarkers and inflammatory cytokines. This approach aims to improve decision-making and predict poor outcomes. In the process of lower respiratory tract infections, the level of procalcitonin (PCT) is intended to guide both the initiation and duration of antibiotic therapy. Additionally, treatment may vary depending on the initial levels of inflammatory biomarkers. Under the influence of pro-inflammatory cytokines (IL-6, G-CSF), CD64 can increase more than tenfold within 4-6 hours. Normally, CD64 expression is low, but it significantly increases within hours when activated by infection. Once the activation subsides, CD64 expression returns to baseline levels within a few days. The summarized data will show correlations between pathogens, their virulence factors, the patient's immune response, and disease outcomes.

Microbiological testing will be conducted when results could influence antimicrobial therapy selection. Sputum microscopy is planned before prescribing antibacterial treatment. Only good-quality sputum samples will be considered for accurate diagnosis. If microscopy reveals poor-quality sputum, further testing will not be pursued. Invasive methods for determining the etiology are intended to be used only when required by pneumonia diagnostic and treatment protocols. The study is planned to be conducted exclusively in specialized hospital units that ensure patient safety. Bronchoscopy, including bronchoalveolar lavage (BAL), is indicated in cases of severe pneumonia and at least one of the following conditions:

* inability to expectorate sputum;
* absence of predominant potential pathogens in sputum culture;
* inadequate response to treatment based on susceptibility of the isolated pathogen;
* isolation of multiple types of Gram-negative rods or fungi in sputum culture;
* suspected superinfection.

In all cases of pneumonia diagnosis, chest X-rays (anteroposterior and/or lateral views) are planned. Infiltrates located in the 2nd, 6th, 9th, and 10th segments may not be visible on the anteroposterior view alone. On the first day of illness, only local changes in the lung pattern-caused by hyperemia, perivascular and peribronchial edema, and infiltration-may be seen. Therefore, chest radiographic examination is planned to be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosed with community-acquired or hospital-acquired pneumonia;
* Provides written informed consent.

Exclusion Criteria:

* Age under 18;
* Inability to provide informed consent;
* Patients with autoimmune diseases;
* Patients with chronic lung diseases such as cystic fibrosis or COPD;
* Contraindications to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult hospitalized patients diagnosed with community-acquired or hospital-acquired pneumonia who meet the inclusion criteria and consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Correlation between inflammatory biomarkers and ICU admission rates | Up to 30 days from enrollment
  Measurement of serum levels of CD64 (index), presepsin (pg/ml), and IL-6 (pg/ml) using a Luminex multiplex assay in patients with community-acquired or hospital-acquired pneumonia and evaluation of their correlation with ICU admission (Incidence of cases/100000 inhabitants).
Correlation between inflammatory biomarkers and hospitalization length | Up to 30 days from enrollment
  Measurement of serum levels of CD64 (index), presepsin (pg/ml), and IL-6 (pg/ml) using a Luminex multiplex assay in patients with community-acquired or hospital-acquired pneumonia and evaluation of their correlation with hospitalization (days).
Correlation between inflammatory markers and a 30-day mortality rate | Up to 30 days from enrollment
  Measurement of serum levels of CD64 (index), presepsin (pg/ml), and IL-6 (pg/ml) using a Luminex multiplex assay in patients with community-acquired or hospital-acquired pneumonia and evaluation of their correlation with 30 day mortality rates (Incidence of cases / 100000 inhabitants)

SECONDARY OUTCOMES:
Measurement of CD64 expression | Within 30 days of enrollment
  Measurement of serum levels of CD64 (index).
Measurement of inflammatory biomarkers | Within 30 days of enrollment
  Measurement of serum levels of presepsin (pg/ml), and IL-6 (pg/ml) in patients

CONTACTS AND LOCATIONS:
Overall Officials: Astra Vitkauskiene, prof. dr., MD, PhD, Study Director — Lithuanian University of Health Sciences
Locations (1):
- Department of Laboratory Medicine, Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including all IPD collected throughout the trial, clinical and biomarker results, will be made available upon reasonable request for scientific research purposes, only IPD used in the results publication. Data will be shared under data use agreements that ensure participant confidentiality.
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: From May 2025 until the End of the Study
Access Criteria: IPD and supporting information will be accesible only to the Investigators using special encrypted cloud database with two-factor authentication and from enlisted secure IP adresses.